CLINICAL TRIAL: NCT04507594
Title: Measurement of Diaphragmatic Dysfunction in Patients Undergoing Thoracic Resection Surgery for Lung- or Esophageal Cancer
Brief Title: Measurement of Diaphragmatic Dysfunction After Thoracic Surgery
Status: Completed | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Peter Juhl-Olsen, Associate Professor, Aarhus University Hospital
Organization: University of Aarhus (Other)
Other Study IDs: DiaphragmaticDysfunction
Record Dates: First submitted 2020-08-06; First posted 2020-08-11 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Diaphragm Injury; Phrenic Nerve Paralysis; Thoracic Cancer; Postoperative Complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing Thoracic Surgery
  Interventions: Procedure: Lung lobectomy OR esophagus cancer resection

INTERVENTIONS:
Procedure: Lung lobectomy OR esophagus cancer resection — Lunge lobectomy (total) Resection of esophagus cancer

SUMMARY:
This study aims to measure diaphragmatic dysfunction with ultrasonography and nerve stimulation of the phrenicus nerve, in patients undergoing thoracic surgery for lung and esophageal cancer, and correlate measures of diaphramatic function to clinical postoperative endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled thoracic resection Surgery for lung- or esophagus cancer. For lung cancer patients, at least one lung lobe has to scheduled for resection

Exclusion Criteria:

* Known Diaphragmatic Dysfunction
* Neuromuscular Disease
* Pleural Effusion > 1cm
* Pneumothorax
* Known Phrenic Nerve Palsy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for resection surgeries for either lung or esophagus cancer.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-08-06 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Change in excursion of the diaphragm | Prior to surgery to 14 days after surgery
  Ultrasonographic measure with M-mode of Diaphragmatic Excursion on right hemidiaphragm

SECONDARY OUTCOMES:
Ultrasonographic measure of the difference in Intrathoracic Area | Prior to surgery to 14 days after surgery
  Intrathoracic Area is measured at inspiration and expiration to calculate the difference in Intrathoracic Area during breathing
Change in Diaphragmatic Thickening Fraction | Prior to surgery to 14 days after surgery
  Ultrasonographic measurement
Change in Intercostal Muscle Thickening Fraction | Prior to surgery to 14 days after surgery
  Ultrasonographic measurement
Change in forced expired volume within the first second (FEV1) | Prior to surgery to 14 days after surgery
  Spirometry
Change in forced vital capacity (FEV) | Prior to surgery to 14 days after surgery
  Spirometry
Change in peak flow | Prior to surgery to 14 days after surgery
  Spirometry
Change in Electromyographic measure of Maximal Diaphragmatic Response after stimulating the phrenic nerve | Prior to surgery to 14 days after surgery
Change in Electromyographic measure of Latency of Diaphragmatic Response after stimulating the phrenic nerve | Prior to surgery to 14 days after surgery
Change in 6 Minutes Walk Test | Prior to surgery to 14 days after surgery
  Maximum Walking Distance within 6 minutes
Change in visual analogue scale score | Prior to surgery to 14 days after surgery
  Scoring system for subjective sensation of pain ranging from 0 to 10. Higher numbers signify higher pain sensations
Accumulated Opiod Use after Surgery | Prior to surgery to 14 days after surgery
  Morphine equivalents
Postoperative Pulmonary Complications | Prior to surgery to 30 days after surgery
  Comprising:
  1. Pneumonia
  2. Atelectasis
  3. Bronchospasm
  4. Hypoxemia
  5. Severe Hypoxemia
  6. Pleural Effusion 1 > cm
  7. Pneumothorax
  8. CPAP or NIV required after 1. postoperative day
Admission days at the Intensive Care Unit after Surgery | Prior to surgery to 60 days after surgery
Number of Admissions after Discharge from the Surgical Department | Prior to surgery to 60 days after surgery
Accumulated Admission Days at any Hospital | Prior to surgery to 60 days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anaesthesiology and Intensive Care East Section, Aarhus University Hospital, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Norskov J, Skaarup SH, Bendixen M, Tankisi H, Morkved AL, Juhl-Olsen P. Diaphragmatic dysfunction is associated with postoperative pulmonary complications and phrenic nerve paresis in patients undergoing thoracic surgery. J Anesth. 2024 Jun;38(3):386-397. doi: 10.1007/s00540-024-03325-5. Epub 2024 Mar 28. PMID 38546897